CLINICAL TRIAL: NCT05528328
Title: Post-surgical Scars After the Use of CACIPLIQ20: A Randomized, Double-blind, Placebo -Controlled Trial
Brief Title: Post-surgical Scars After the Use of CACIPLIQ20
Acronym: MATRISCAR
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Organ, Tissue, Regeneration, Repair and Replacement (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-A00833-40
Record Dates: First submitted 2022-08-29; First posted 2022-09-06 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Scars
Keywords: mammoplasty
MeSH Terms: conditions — Cicatrix | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: This is a prospective double-blinded placebo self-controlled trial. 50 female patients undergoing bilateral mammoplasty for breast hypertrophy will be included.CACIPLIQ20® will be administered topically on the vertical and peri-areolar incisions of one breast for 5 minutes, after subcutaneous plans suture and just before final skin suture. The placebo will be administered in the same manner on the contralateral breast. As a result, each patient will receive both CACIPLIQ20® and placebo, thus reducing the interpersonal variability with a self-controlled design.The treatment assignment for each breast will be randomized.The patient, investigator and adjudication committee will be blinded during the whole study, until all assessments have been performed.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study is a double-blind study. Each product, CACIPLIQ20® or placebo, will be supplied in vials having the same appearance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CACIPLIQ20® (Active Comparator): CACIPLIQ20® is a medical device used for the treatment of chronic skin ulcers, and contains a molecule belonging to the family of ReGeneraTing Agents (RGTA®). CACIPLIQ20® will be administered topically on the vertical and peri-areolar incisions of one breast for 5 minutes, after subcutaneous plans suture and just before final skin suture.
  Interventions: Device: CACIPLIQ20®
- placebo (Placebo Comparator): The placebo solution (saline solution) will be administered on the contralateral side.
  Interventions: Drug: Placebo (saline solution)

INTERVENTIONS:
Device: CACIPLIQ20® — CACIPLIQ20®
  Arms: CACIPLIQ20®
Drug: Placebo (saline solution) — Placebo (saline solution) administered in identic al vials
  Arms: placebo

SUMMARY:
Following surgical procedures or injury, cutaneous scars can develop due to production of collagen-rich connective tissue. These scars may be accompanied by redness, itching, pain, and restricted mobility of the skin. Typically, after a few weeks, the scar matures, becoming lighter and narrower, although full maturation of a scar may take up to 2 years. In some cases, however, cutaneous scars can be unsightly or can even become hyper- trophic or result in keloids.

Preventing pathological scarring is much easier than treating scars later and should be started as early as possible after the injury or surgery.

CACIPLIQ20® is a medical device used for the treatment of chronic skin ulcers, and contains a molecule belonging to the family of ReGeneraTing Agents (RGTA®). RGTA®s are biodegradable polymers that mimic the action of heparan sulfates found in the extracellular matrix of injured tissues. RGTA® accelerates tissue healing in various animal models, by stabilizing and protecting heparin-binding growth factors (HBGFs) and matrix proteins. In addition to its effects on hard-to-heal chronic wounds, CACIPLIQ20® was found to improve acute wound healing in pre-clinical models and in several case reports and controlled clinical studies. A first open label-controlled study showed that the topical application of RGTA® improved skin healing in mammoplasty patients and notably reduced oedema and pain in patients who had undergone centrofacial lift surgery compared to untreated patients. Results from this first study were confirmed in a double-blind placebo self-controlled trial conducted in two medical institutions in China involving 71 patients. The Chinese study showed that a single application of CACIPLIQ20® significantly improved scar healing quality at 14 days as well as scar symptoms including pain, swelling and exudate. The aim of the MATRISCAR study is to confirm the previous results in a double-blind, placebo-controlled randomized clinical trial.

DETAILED DESCRIPTION:
MATRISCAR is a double-blind, placebo-controlled, self-controlled, randomized clinical trial.

The main objective of this pivotal trial is to assess the superiority of a single application of CACIPLIQ20® over placebo on the clinical outcomes of the scars at 24 weeks. The primary endpoint will be the overall opinion on the appearance of the scar at 24 weeks, using the global scar comparison scale, centrally performed by an adjudication committee.

It is planned to include 50 female patients undergoing bilateral mammoplasty for breast hypertrophy, from 3 centers in France. Each subject's participation duration in the study is estimated to be 6 months. The enrolment period is estimated to be 8 to 10 months.

The targeted mammoplasties consist in the surgical reduction of both breasts volume, resulting in almost symmetrical scars. Surgical incisions of the bilateral breast reduction will be sutured according to local standard procedures. CACIPLIQ20® will be administered topically on the vertical and peri-areolar incisions of one breast for 5 minutes, after subcutaneous plans suture and just before final skin suture. The placebo will be administered in the same manner on the contralateral breast. As a result, each patient will receive both CACIPLIQ20® and placebo, thus reducing the interpersonal variability with a self-controlled design.

Standardized two-dimensional (2D) photographs of each scar will be collected at 4, 12 and 24 weeks by the investigator, as well as other clinical outcomes. The scars photographs of each patient at each visit will be placed side by side (i.e. 2 photos per patient/visit), for a centralized evaluation by an adjudication committee.

The treatment assignment for each breast will be randomized at treatment labelling. Treatments (active and placebo) will be dispensed in identical vials of 5 ml identified by treatment numbers and letters (R for the right breast, L for the left breast). The patient, investigator and adjudication committee will be blinded during the whole study, until all assessments have been performed. The independent monitor will ensure blinding is respected.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for bilateral breast reduction (>300 g by breast) using the conventional superior pedicle technique with inverted-T scars
2. Age between 18 and 85 years
3. Patients having received a full written and oral information about study conduct and objectives
4. Patients who can and are willing to be followed by the study investigator for the duration of the study
5. Patients benefiting from a valid health insurance or social security coverage

Exclusion Criteria:

1. Female patients who are pregnant, or lactating
2. Patients with, according to investigator's opinion, a very poor life expectancy
3. Patients intolerant to one of the study device components or to heparinoids
4. Any scar treatment other than the standard of care
5. Previous breast surgery
6. Current malignancy

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
differential appearance of the treated and untreated (placebo) scars at 24 weeks, using the global scar comparison scale assessed by a blinded adjudication committee composed of 3 experts. | Up to 24 weeks (the primary endpoint will be judged at 24 weeks)
  The global scar comparison scale (GSCS), ranging to -100 to +100, indicates by how much one of the scars has a better appearance than the contralateral scar. A positive score means that the CACIPLIQ side is improved and higher values mean higher improvement compared to the contralateral side.

SECONDARY OUTCOMES:
Proportion, of scars improved by at least 30% at 12 weeks and 24 weeks based on the global scar comparison scale | up to 24 weeks (12 and 24 weeks)
  The global scar comparison scale, ranging to -100 to +100, indicates by how much one of the scars has a better appearance than the contralateral scar. Higher scores mean higher improvement on the treated side.
Pruritus assessed by a Visual Analogue Scale (Pruritus VAS) | Up to 4 weeks
  This scale consists of a 10cm long line and a single question. It is most commonly used in clinical trials for measuring itch intensity and features high reliability and concurrent validity. The left end point represents "no itch" and the right end point the "worst imaginable itch". The higher the score (from 0 to 10), the higher the pruritus is.
Mean observer POSAS (Patient and Observer Scar Assessment Scale) scale | At 24 weeks
  The POSAS is a reliable and valid scar assessment scale that measures scar quality from two perspectives: the patient and the clinician. The POSAS measures scar quality in all types of scars by evaluating visual (e.g. color), tactile (e.g. pliability) and sensory (e.g. itch) characteristics of the scar. The total score ranges from 7 to 70. Higher scores are associated with poor scar outcome .
Mean patient POSAS (Patient and Observer Scar Assessment Scale) scale | At 24 weeks
  The POSAS is a reliable and valid scar assessment scale that measures scar quality from two perspectives: the patient and the clinician. The POSAS measures scar quality in all types of scars by evaluating visual (e.g. color), tactile (e.g. pliability) and sensory (e.g. itch) characteristics of the scar. The total score ranges from 7 to 70. Higher scores are associated with poor scar outcome .
Pain assessed by a Visual Analogue Scale (Pain VAS) | Up to 4 weeks
  The visual analogue scale (VAS) is a tool widely used to measure pain. A patient is asked to indicate his/her perceived pain intensity (most commonly) along a 100 mm horizontal line, and this rating is then measured from the left edge (=VAS score). The score ranges from 0 (no pain) to 100 (severe intolerable pain). Higher scores are associated with higher pain intensity.
Rate of adverse events (AEs) | up to 24 weeks
  including serious and non-serious AEs, anticipated or unanticipated AEs, related to CACIPLIQ20® use, according to investigators' opinion
Rate of device deficiencies (DDs) | up to 24 weeks
  Device deficiencies related to CACIPLIQ20® use, according to investigators' opinion

CONTACTS AND LOCATIONS:
Overall Officials: Gilbert Zakine, Principal Investigator — Clinique Turin
Locations (2):
- France (2):
  - CHU Brest, Brest, Brittany Region
  - Clinique Turin, Paris, Île-de-France Region